CLINICAL TRIAL: NCT06155188
Title: A Novel Post-transplant Regimen of PT/FLU+CY for Selectively Promoting Unrelated Cord Blood Engraftment in Haploidentical-cord Transplantation in Childhood Leukemia: a Single-arm, Multi-center Trial
Brief Title: Post-transplant PT/FLU+CY Promotes Unrelated Cord Blood Engraftment in Haplo-cord Setting in Childhood Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-229
Record Dates: First submitted 2023-11-13; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Leukemia; Stem Cell Transplant; Cord Blood
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PT/FLU+CY (Experimental): The group consisted of fludarabine (40mg/m2, day-5 to day-3 and day+3, day+4), busulfan (100mg/m2, day-6 to day-3), haplo-PBSC (day0), cyclophosphamide (50mg/kg, day+3, day+4) , and UCB (day+6)
  Interventions: Procedure: applying of FLU+CY post-HSCT

INTERVENTIONS:
Procedure: applying of FLU+CY post-HSCT — The conditioning regimen (PT-Cy/Flu group) consisted of fludarabine (40mg/m2, d-5 to d-3 and d+3, d+4), busulfan (100mg/m2, d-6 to d-3), haplo-PBSC (d0), PTCy (50mg/kg, d+3, d+4) and UCB (d+6).

SUMMARY:
To determine if the novel regimen of PT/FLU+CY promotes cord blood engraftment in children's leukemia HSCT cohort

DETAILED DESCRIPTION:
PTCy is a well-established haploidentical transplant regimen strategy. Moreover, unrelated cord blood (UCB) plays a critical role in the effects of GVL. However, the engraftment of grafts is unpredictable in the setting of a haplo-cord subsequent transplant. Therefore, applying a novel post-transplant regimen of PT/CY+FLU may selectively promote UCB engraftment in the setting of haplo-cord transplant.

ELIGIBILITY:
Inclusion Criteria:

* children acute leukemia

Exclusion Criteria:

* MODS

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
rate of UCB engraftment | initiate STR detection from day+15 thereafter weekly up to 1 year post-HSCT
  evaluate the regimen if it promotes UCB engraftment
rate of leukemia free survival | 3 years post-HSCT
  determine the leukemia status post-HSCT
rate of overall survival | 3 years post-HSCT
  determine the overall survival status post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqin Feng, MD, Principal Investigator — Department of Pediatrics, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China